CLINICAL TRIAL: NCT06853184
Title: Phase 2, Randomized, Open-label, Active Comparator, Dose-ranging Study Evaluating the Efficacy and Safety of Artesunate for Injection in Combination With Ganciclovir or Valganciclovir for the Treatment of Cytomegalovirus Infection in Solid Organ Transplant Recipients
Brief Title: Study Evaluating the Efficacy and Safety of Artesunate
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amivas Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVAS-CMV-01
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: CMV Infection
Keywords: CMV infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Artesunate; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Artesunate (Experimental): Low Dose Artesunate: 2.4 mg/kg IV artesunate once daily for 14 days + GCV or VGCV and SOC per local institutional practices
  Interventions: Drug: Artesunate
- High Dose Artesunate (Experimental): High Dose Artesunate: 4.8 mg/kg IV artesunate once daily for 14 days + GCV or VGCV and SOC per local institutional practices
  Interventions: Drug: Artesunate
- Standard Treatment Ganciclovir (Active Comparator): Standard Treatment Ganciclovir: GCV or VGCV and SOC per local institutional practices
  Interventions: Drug: Ganciclovir (GCV)

INTERVENTIONS:
Drug: Artesunate — Low Dose Artesunate: 2.4 mg/kg IV artesunate once daily for 14 days + GCV or VGCV and SOC per local institutional practices High Dose Artesunate: 4.8 mg/kg IV artesunate once daily for 14 days + GCV or VGCV and SOC per local institutional practices
  Arms: High Dose Artesunate; Low Dose Artesunate
Drug: Ganciclovir (GCV) — Standard Treatment Ganciclovir: GCV or VGCV and SOC per local institutional practices
  Arms: Standard Treatment Ganciclovir

SUMMARY:
This study is a randomized, open-label, active comparator-controlled, dose-ranging trial of the efficacy and safety of IV artesunate in combination with IV GCV or oral VGCV and SOC treatment compared to GCV or VGCV monotherapy and SOC treatment in SOT recipients with clinically significant CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Recipient of a solid organ transplant (kidney, lung, heart, or liver)
* Have a documented CMV infection
* Have CMV DNAemia
* Require IV GCV or oral VGCV
* Be washed out from any anti-CMV antiviral drugs
* Have all the following results as part of screening laboratory assessments
* Have life expectancy of ≥ 12 weeks
* Be willing and have an understanding and ability to fully comply with the study
* If female use birth control

Exclusion Criteria:

* Have taken IV GCV or oral VGC daily for >8 days
* Have refractory CMV infection or disease
* Have CMV antiviral drug resistance
* Have a known hypersensitivity to artesunate, GCV, or VGCV
* Pregnant (or expecting to conceive) or nursing
* Have severe liver disease
* Require ongoing treatment with or an anticipated need for treatment with drugs with known interactions with artesunate or GCV
* Taking any another investigational drug with anti-CMV activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of cytomegalovirus (CMV) DNAemia | 28 days
  Determine if Artesunate for Injection (intravenous [IV] artesunate) when administered in combination with IV Ganciclovir (GCV) and/or oral valganciclovir (VGCV) and standard of care (SOC) treatment impacts change of cytomegalovirus (CMV) DNAemia compared with those who only received GCV or VGCV and SOC treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Westmead Hospital, Westmead
  - Princess Alexandra Hospital, Woolloongabba

IPD SHARING:
Plan to Share IPD: No